CLINICAL TRIAL: NCT05111977
Title: A Neurocomputational Assay of Gastrointestinal Interoception in Anorexia Nervosa
Brief Title: Gastrointestinal Interoception in Anorexia Nervosa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: R01MH127225 (NIH)
Record Dates: First submitted 2021-10-19; First posted 2021-11-08 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Anorexia Nervosa
Keywords: Interoception
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Capsule stimulation (Experimental): Participants in this arm will receive gastric stimulation via the Vibrant capsule
  Interventions: Device: Vibrant capsule
- Placebo stimulation (Placebo Comparator): Participants in this arm will receive no gastric stimulation via a placebo capsule
  Interventions: Device: Vibrant capsule

INTERVENTIONS:
Device: Vibrant capsule — A capsule delivering mechanical vibrations

SUMMARY:
Anorexia nervosa (AN) has among the highest mortality rate of any psychiatric illness, yet we have a poor understanding of the biological causes of this disorder. In this study, we use a novel mechanosensory intervention to examine the basic question of whether individuals with AN have abnormal "gut sensations" and whether such indicators are associated with adverse consequences from the disorder.

ELIGIBILITY:
Inclusion Criteria:

HC Inclusion criteria:

i. Body mass index ≥ 18.5. ii. Females, ages 15 to 40 years iii. Women of childbearing age: a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study.

iv. Independently ambulatory v. Possession of a smartphone with data plan vi. English proficiency vii. Willingness and ability to participate in study procedures viii. Provision of signed and dated informed consent form

AN Inclusion criteria:

i. Primary clinical diagnosis of anorexia nervosa as defined by Laureate Eating Disorders Program ii. Body mass index ≥ 18.5. iii. Transitioned from acute clinical status rating to residential clinical status or partial/intensive outpatient clinical status rating iv. No new medication prescription in the week prior to study randomization, Must be on a stable dose of medication for at least 1 week.

v. Females, ages 15 to 40 years vi. Women of childbearing age: a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study.

vii. Independently ambulatory viii. Possession of a smartphone with data plan ix. English proficiency x. Willingness and ability to participate in study procedures xi. Provision of signed and dated informed consent form

Exclusion Criteria:

HC Exclusion criteria:

i. Current diagnosis of a psychiatric disorder per the MINI International Diagnostic Interview

ii. Taking any psychotropic medication

iii. Active suicidal ideation with intent or plan

iv. Active cutting or skin lacerating behaviors

v. Active purging behaviors (specifically, self-induced vomiting), and/or a history of severe self-induced vomiting

vi. Pregnancy as defined by a urine screen during screening, and confirmed during each stimulation visit, and must not be lactating

vii. History of significant gastrointestinal disorder, including any form of inflammatory bowel disease or gastrointestinal malignancy (celiac disease is accepted if the subject has been treated and is in remission)

viii. History of complicated/obstructive diverticular disease

ix. Clinical evidence of significant gastroparesis

x. Diagnosis of mega-rectum or colon, congenital anorectal malformation, or clinically significant rectocele or rectal prolapse

xi. History of intestinal or colonic obstruction, or suspected intestinal obstruction

xii. History of intestinal resection (with an exception for appendectomy, cholecystectomy and inguinal hernia repair), history of bariatric surgery or evidence of any structural abnormality of the gastrointestinal tract that might affect transit

xiii. History of Zenker's diverticulum, dysphagia, Barrett's esophagus, esophageal stricture or achalasia, transesophageal fistula, or eosinophilic esophagitis.

xiv. Clinical evidence (as judged by the investigator) of respiratory, cardiovascular, renal, hepatic, biliary, endocrine, or neurologic disease

xv. Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs): chronic use is defined as taking full dose NSAIDs more than three times a week for at least six months. Subjects on cardiac doses of aspirin may be enrolled in the study

xvi. Cardiac pacemaker, implantable cardioverter defibrillator, implantable infusion device, or gastric electrical stimulator

xxv. Orthostatic hypotension (defined as a drop of ≥ 20 mm Hg in systolic BP or a drop of ≥ 10 mm Hg in diastolic BP when measured shortly after transitioning from lying down to standing)

xxvi. Any other condition which in the opinion of the investigator may adversely affect the safety of the subject or would limit the subject's ability to complete the study

xxvii. No smartphone/computer or limited access to a smartphone/computer

xxviii. Regular use of any of the following medications or procedures: Medications that may substantially affect intestinal motility, prokinetics at high doses (metoclopramide, erythromycin, senna, prucalopride), anti-Parkinsonian medications, opiates, opioids, calcium-channel blockers, enemas

xxix. History of a GI bleed within the last 3 months

xxx. Pelvic floor dysfunction/defecatory disorder, based on subject history

xxxi. Planning to undergo MRI during study time frame

xxxii. Any known allergy to soybean or beeswax or Calcium Carbonate

xxxiii. Bradycardia less than 40 beats per minute

xxxiv. Pain Disorder

AN Exclusion criteria:

i. Active suicidal ideation with intent or plan

ii. Active cutting or skin lacerating behaviors

iii. Active purging behviors (specifically, self-induced vomiting), and/or a history of severe self-induced vomiting

iv. Pregnancy as defined by a urine screen during screening, and confirmed during each stimulation visit, and must not be lactating

v. History of significant gastrointestinal disorder, including any form of inflammatory bowel disease or gastrointestinal malignancy (celiac disease is accepted if the subject has been treated and is in remission)

vi. History of complicated/obstructive diverticular disease

vii. Clinical evidence of significant gastroparesis

viii. Diagnosis of mega-rectum or colon, congenital anorectal malformation, or clinically significant rectocele or rectal prolapse

ix. History of intestinal or colonic obstruction, or suspected intestinal obstruction

x. History of intestinal resection (with an exception for appendectomy, cholecystectomy and inguinal hernia repair), history of bariatric surgery or evidence of any structural abnormality of the gastrointestinal tract that might affect transit

xi. History of Zenker's diverticulum, dysphagia, Barrett's esophagus, esophageal stricture or achalasia, transesophageal fistula, or eosinophilic esophagitis.

xii. Clinical evidence (as judged by the investigator) of respiratory, cardiovascular, renal, hepatic, biliary, endocrine, or neurologic disease

xiii. Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs): chronic use is defined as taking full dose NSAIDs more than three times a week for at least six months. Subjects on cardiac doses of aspirin may be enrolled in the study

xiv. Cardiac pacemaker, implantable cardioverter defibrillator, implantable infusion device, or gastric electrical stimulator

xv. Orthostatic hypotension (defined as a drop of ≥ 20 mm Hg in systolic BP or a drop of ≥ 10 mm Hg in diastolic BP when measured shortly after transitioning from lying down to standing)

xvi. Any other condition which in the opinion of the investigator may adversely affect the safety of the subject or would limit the subject's ability to complete the study

xvii. No smartphone/computer or limited access to a smartphone/computer

xviii. Regular use of any of the following medications or procedures: Medications that may substantially affect intestinal motility, prokinetics at high doses (metoclopramide, erythromycin, senna, prucalopride), anti-Parkinsonian medications, opiates, opioids, calcium-channel blockers, enemas

xix. History of GI bleed within the last 3 months

xx. Pelvic floor dysfunction/defecatory disorder, based on subject history

xxi. Planning to undergo MRI during study time frame

xxii. Any known allergy to soybean or beeswax, or Calcium Carbonate

xxiii. Bradycardia less than 40 beats per minute

xxiv. Pain Disorder

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Interoceptive precision | At baseline
  Interoceptive sensory precision
Interoceptive prior | At baseline
  Interoceptive prior expectaiton
Learning rate | At baseline
  Interoceptive learning rate
Evoked response potential | At baseline
  Electroencephalogram (EEG) evoked response amplitude within 700 millisecond period following vibration onset
Electrogastrogram | At baseline
  Stomach electrogastrogram (EGG) power in bradygastria, normogastria, tachygastria and total power bands

SECONDARY OUTCOMES:
Normalized A prime | At baseline
  Signal detection accuracy measure
Illness status | At 1 month, 3 month, and 6 month follow-up
  Relapse, remission, or recovery status

CONTACTS AND LOCATIONS:
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
We will upload the collected data via the NIMH Data Archive (NDA) data repository.
Time Frame: Data will be available approximately one year after the end of the study period.